CLINICAL TRIAL: NCT06438133
Title: Digital Supported Compression Bandaging in Patients With Chronic Edema in the Lower Limbs - Assessment of Measurement Properties of a Novel Sensor
Brief Title: Digital Supported Compression Bandaging in Patients With Chronic Edema in the Lower Limbs
Acronym: CIMON
Status: Completed | Type: Observational
Sponsor: Carsten Bogh Juhl (Other)
Collaborators: Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other); Odense University Hospital (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor-Investigator, Carsten Bogh Juhl, Professor, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Other Study IDs: CIMON
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Compression; Vein; Venous Insufficiency; Lymphedema of Leg; Digital Technology
Keywords: Compression therapy; Compression bandaging; Chronic edema; Psychometrics
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic edema of the lower limbs: Patients with chronic edema of the lower limbs referred to compression bandaging in a hospital setting.
  Interventions: Other: CIMON; Other: Sens Motion

INTERVENTIONS:
Other: CIMON — The sensor assess changes in the circumference of the limb and will be applied to the lower limb before compression bandaging is applied.
Other: Sens Motion — The sensor assess physical activity and the amount of time spent at rest, standing, walking, running and count steps.

SUMMARY:
Patients with chronic edema of the lower limb referred to compression bandaging in a hospital setting will be invited to participate in the validation study of a novel sensor (CIMON), which have been developed for assessing the effect of compression bandaging. Participants will have the sensor applied to the lower limb before initiation of compression bandaging and will receive usual compression treatment according to severity of the edema and usual practice at the treatment site. Duration of participation is 14 days.

DETAILED DESCRIPTION:
The CIMON sensor is developed with the purpose of monitoring the effectiveness of compression bandaging (CB) in patients with chronic edema by application to the widest circumference of the calf. CIMON measures the difference in capacitance by stretching the circumferential sensor. Data from the sensor is transferred by Bluetooth technology to a secured webserver, where healthcare professionals can monitor the effect of compression bandaging.

The study aims to assess the psychometric properties of the CIMON (reliability, validity and responsiveness) and assess the correlation between edema reduction and physical activity during compression bandaging.

ELIGIBILITY:
Inclusion Criteria:

* Chronic edema of the lower limb
* Referred to compression bandaging
* Circumference of widest point of the lower leg between 35-75 cm

Exclusion Criteria:

* Wounds at the lower leg (at the widest circumference of the lower leg)
* Acute deep venous thrombosis in the leg
* Untreated cellulitis
* Severe heart- or kidneyfailure
* Severe peripheral neuropathy in the lower limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic edema of the lower limbs referred to compression bandaging in a hospital setting.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Edema reduction | 14 days
  Assessed by Cimon sensor (in capacitans, pF)

SECONDARY OUTCOMES:
Edema reduction | 14 days
  Assessed by tape measurement (in cm), converted to volume by formula of truncated cone
Edema reduction | 14 days
  Assessed by perometry (in ml)
Edema reduction | 14 days
  Assessed by Dual energy X-ray Absorptiometry (in kg)
Symptoms related to chronic edema | 14 days
  Self-reported pain, tension and heaviness
Physical Activity (PA) | 14 days
  Assessed by Sens Motion sensor (PA by sedentary time, low+moderate and high intensity in minutes)
Adverse events | 14 days
  Any adverse events related to compression bandaging and the application of sensors

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bogh Juhl, Professor, Study Chair — Herlev and Gentofte Hospital
Locations (5):
- Denmark (5):
  - Department of Dermatology, Frederiksberg Bispebjerg Hospital, Bispebjerg, Capital Region
  - Department of Physiotherapy and Occupational Therapy, Rigshospitalet, Copenhagen, Capital Region
  - Department of Physiotherapy and Occupational Therapy, Herlev and Gentofte Hospital, Herlev, Capital Region
  - Department of Physiotherapy and Occupational Therapy, Amager Hvidovre Hospital, Hvidovre, Capital Region
  - Department of Oncology, Unit of Lymphedema care, Odense University Hospital Svendborg, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No